CLINICAL TRIAL: NCT01231308
Title: Roux-en-Y-Gastric Bypass (RYGB) Versus Lifestyle Modification Plus Medical Therapy in the Treatment of Type 2 Diabetes in Overweight-to-Moderately Obese Patients: A Randomized Clinical Trial
Brief Title: Roux-en-Y-Gastric Bypass vs. Lifestyle Modification and Medical Therapy in the Treatment of Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1002010906
Record Dates: First submitted 2010-10-27; First posted 2010-11-01 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle modification (Active Comparator): Intensive nutritional/exercise counseling for weight loss by lifestyle modification in addition to optimum medical treatment.
  Interventions: Behavioral: Intensive lifestyle modification and Optimal medical Therapy
- Roux-en-Y-Gastric Bypass (Experimental): A laparoscopic gastric bypass will be performed in the treatment of type 2 diabetes in Overweight-to-Moderately Obese Patients
  Interventions: Procedure: Roux-en-Y-Gastric Bypass

INTERVENTIONS:
Procedure: Roux-en-Y-Gastric Bypass — Standard laparoscopic gastric bypass. Preoperative preparation will include antibiotic prophylaxis given less than 60 minutes prior to making the first incision. Under general anesthesia with endotracheal intubation, a laparoscopic gastric bypass will be performed in the usual fashion.
  Arms: Roux-en-Y-Gastric Bypass
Behavioral: Intensive lifestyle modification and Optimal medical Therapy — Very low calorie diet consisting of 5 feedings: 2 liquid meal replacements, 2 low-calorie snacks, and 1 small meal of known caloric content. After 10% weight loss is achieved, the subjects will received individualized nutrition sessions beginning bi-weekly but extending time intervals as the weight loss progresses.
  Arms: Lifestyle modification

SUMMARY:
The study is aimed to compare: Laparoscopic Roux-en-Y-Gastric Bypass (RYGB) + optimal medical therapy versus Intensive lifestyle modification and optimal medical therapy in the treatment of type 2 diabetes in overweight-to-moderately obese patients (BMI: 28-34kg/m2; the lower BMI cut-off will be 26kg/m2 in patients of Asian descent).

This is a single center, prospective randomized study. The study at the Weill College Medical College Diabetes Surgery Center. This study is intended to be a pilot investigation whose results can inform clinicians and researchers for future larger or multi-site trials of diabetes surgery. This study will also be used for the definition of a "core" protocol for independent randomized clinical trials to be carried out at various centers participating in a multinational consortium.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes by any of the following:

   * A fasting plasma glucose > 126 mg/dl confirmed on repeated testing
   * 2 hour plasma glucose > 200mg/dl during a 75 gram oral glucose tolerance test
   * HbA1c >6.5%
2. A normal or high C-peptide level (> 0.9 ng/ml) to exclude type 1 diabetes and insulin deficient type 2 diabetes
3. Negative AntiGAD 65 Antibodies
4. Body mass index (BMI) between 28 and 35 kg/m2 ( > 27.6 kg/m2 and < 34.5 kg/m2 ) that reflect a condition of overweight to moderate obesity.

   In consideration of the evidence that the associations between BMI, percentage of body fat, and CV risk differ across populations, and that the proportion of Asian people with a high risk of type 2 diabetes and cardiovascular disease is substantial at BMI's lower than the existing WHO cut-off point for overweight (= 25 kg/m2) (source: WHO Expert consultation. Lancet. 2004 Jan 10;363(9403):157-63), the lower BMI cut-off for inclusion in this study will be 26kg/m2 for patients of Asian descent.
5. No contraindications for surgery or General Anesthesia as determined by a multidisciplinary team (surgeon, endocrinologist/internist, cardiologist, nutritionist)
6. . Between 21 and 65 years of age
7. . Able to provide informed consent
8. . If a female with reproductive potential, agreement to use a reliable method of birth control for 2 years following surgery (Barrier, birth control, patch).

   This precaution is necessary to prevent potential complications of pregnancy due to possible nutritional deficiencies in the period of more intense weight loss after surgery. On the other hand, this precaution will avoid erratic weight/glucose tolerance changes of pregnancy effecting results.
9. Have valid health insurance

Exclusion Criteria:

1. Diagnosis of diabetes more than 15 years (to exclude pts with significant decline in pancreatic function from long-standing diabetes)
2. Insulin therapy for more than 12 years
3. HbA1c higher than 10%
4. Diagnosis of type 1 diabetes
5. Enrolled in another clinical study which involves an investigational drug
6. Major psychological disorders
7. Pregnancy (all female patients will have serum beta hCG) or planned pregnancy within two years of entry into the study or unwilling to use reliable contraceptive method
8. Previous gastric or esophageal surgery
9. Immunosuppressive drugs including corticosteroids
10. Coagulopathy (INR > 1.5 or platelets < 50,000/μl)
11. Anemia (Hb < 10.0 g/dl)
12. Any contraindication to laparoscopic gastric bypass or medical diabetes therapy
13. A severe concurrent illness likely to limit life (e.g. cancer) or requiring extensive systemic treatment (e.g. ulcerative colitis)
14. A significant malabsorptive or gastrointestinal disorder (e.g. pancreatic insufficiency, Celiac sprue, or Crohn's disease)
15. Significant proteinuria (> 250 mg/dl)
16. Severe neuropathy or clinical diagnosis of gastropathy (early satiety, nausea, vomiting, constipation alternating with diarrhea)
17. Myocardial infarction in the previous year, current angina or heart failure

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
The primary end-point will be the control of hyperglycemia (HbA1c <6.5% + FG<126mg/dl). | Monthly after initiation of study for a minimum of 3 months, and then every monthly until HbA1c is below 7%

SECONDARY OUTCOMES:
Short (2 yrs) and long term (5 yrs.) achievement of 'adequate" glycemic control, mean change in HbA1c from baseline. | Year 2 and year 5

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Rubino, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States